CLINICAL TRIAL: NCT05553418
Title: BD Evolve On-body Injector: Clinical Feasibility and Performance in the Abdomen and Arm
Brief Title: Investigational On-body Injector Clinical Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Becton, Dickinson and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: PHS-20OBI01
Record Dates: First submitted 2022-07-15; First posted 2022-09-23 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Healthy Volunteers
Keywords: On-Body Injector

STUDY DESIGN:
Intervention Model Description: All participants will participate in three (3) study arms, whereby each participant will wear six (6) OBI prototype devices in total: three (3) on the arm and three (3) on the abdomen. A randomization scheme will be provided with the order of study arm + body location (arm/abdomen) + body side (left/right) randomized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "In-Clinic wear first" (Experimental): Participant will wear the devices first during 27 hr in-clinic wear first followed by injection, then a short-term wear period in-clinic followed by injection, and finally at home for 27 hrs followed by injection.
  Interventions: Device: In-clinic wear first
- "Home wear first" (Experimental): Participant will wear the devices at home first with return to clinic for injection, followed by a short-term wear period in-clinic for injection, and finally during a 27hr in-clinic stay for injection
  Interventions: Device: Home wear first

INTERVENTIONS:
Device: In-clinic wear first — Participant will remain in clinic and wear devices adhered on abdomen or arm approximately 27hrs prior to injection
  Arms: "In-Clinic wear first"
Device: Home wear first — Device will be applied to the abdomen or arm to deliver placebo subcutaneously. After device application, participant will go home and return to clinic before delivery.
  Arms: "Home wear first"

SUMMARY:
The purpose of this study is to evaluate the clinical feasibility, performance, safety and acceptability of the On-body Injector (OBI) when applied to the arm or abdomen of healthy volunteers to inject placebo under the skin.

DETAILED DESCRIPTION:
This study is a monocentric, open-label, cross-over, feasibility and exploratory study with no acceptance criteria. Up to 70 healthy volunteers will be enrolled and followed up for 7 weeks at maximum.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult participants ≥ 18 years
* BMI ≥18.5 kg/m2
* Participant willing and able to complete all required study procedures and to provide informed consent

Exclusion Criteria:

* Participant any self-reported existing chronic illness (heart disease, respiratory disease, kidney disease, metabolic diseases etc.).
* Participants with treatment interfering with coagulation, platelet function, or pain perception within 12 hrs of in-clinic visit
* Participants with abdominal or arm skin conditions or treatments that may interfere with planned study treatment
* Participants with acute or chronic hepatitis B or C and/or with known history/positive HIV serology.
* Participants who are pregnant, planning to become pregnant, or are breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2022-09-05 (Actual); Primary Completion 2023-02-08 (Actual); Study Completion 2023-02-08 (Actual)

PRIMARY OUTCOMES:
Device Performance - Dose delivery efficiency | After device removal
  Determined by volume - measured via gravimetric analysis (weighing the device)
Device Performance | From device application until 15-minutes after injection
  Change in adhesive pad adherence - device to skin/device to adhesive pad - determined via adherence scales (Score 0 - 4, whereby 0 is full adherence and 4 is reflecting full detachment)

SECONDARY OUTCOMES:
Additional OBI performance - Injection signal/indicator performance | Before, during and after injection for each applied device; up to 28 hours after application
  Assessed by visual or audible observation from activation to injection end.
Additional OBI performance - Catheter condition | Approximately 15-minutes after device removal
  Catheter bending assessment by grading
Participant Pain | Immediately before device catheter is inserted, after insertion, during wear period, at start of injection, 15 minutes after injection, end of injection and upon removal for each applied device
  100mm Visual Analog Scale (VAS) for pain assessment - describing no pain with 0mm - up to worst possible pain described with 100mm
Participant Acceptability Questionnaires | Device acceptability questionnaire will be completed after device catheter is inserted, at 8 hours and 26 hrs after application, during Injection and upon device removal
  Questionnaires to assess participants' acceptability of the device during wear
Ultrasound Imaging of injection site | Baseline and immediately after procedure for each applied device
  Measure pre- and post-injection tissue thickness
Tissue Effects | Baseline, immediately after procedure, follow up check up to 72 hours after injection in case tissue effects are present
  Assessment of wheal and erythema described via grading 0-4, incidence of bleeding, bruising, induration
Adverse Events | Throughout study completion, an average of 4 week
  Incidence of adverse device effects and procedure related adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Yves Donazzolo, MD, Principal Investigator — Eurofins
Locations (1):
- Eurofins Optimed, Gières, France

IPD SHARING:
Plan to Share IPD: No